CLINICAL TRIAL: NCT04557358
Title: Impact in the Medical Care Among the Rheumatic Diseases Patients in a Tertiary Hospital in México During the COVID-19 Pandemic
Brief Title: Impact in the Medical Care Among the Rheumatic Diseases Patients in a Hospital in México During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Principal Investigator, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-3467
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis; Quality of Life
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatic diseases outpatients: All the rheumatic diseases outpatients from the National Institute of Medical Sciences and Nutrition that will assist their usual medical care posterior of stopped it during the COVID-19 pandemic.
  In order to explore how the patient´s disease activity, patient´s quality of life, and psychopathology will change with the reintegration at medical care, randomization 200 rheumatic diseases outpatients that will respond RAPID-3 (disease activity/disease severity), WHOQOL-BREF instrument (quality of life), DASS-21 instrument (depression and anxiety), IER-R (posttraumatic stress)
  Interventions: Other: COVID-19 survey; Other: RAPID-3; Other: WHOQOL-BREF; Other: DASS-21 instrument (depression and anxiety); Other: IER-R (posttraumatic stress)

INTERVENTIONS:
Other: COVID-19 survey — A questionnaire locally developed to explore access to medical care and to medications, access to communication with their primary rheumatologist, and patients risk perception about COVID-19 disease
Other: RAPID-3 — The instrument measures function, pain, and patient global estimate of status, with correspond to activity disease
Other: WHOQOL-BREF — The instrument measures the patient´s quality of life (4 dimensions: physics, phycological, social, and environment)
Other: DASS-21 instrument (depression and anxiety) — The instrument measures the presence of depression and anxiety
Other: IER-R (posttraumatic stress) — The instrument measures the presence of posttraumatic stress

SUMMARY:
The National Institute of Medical Sciences and Nutrition is a national reference center for rheumatic diseases that belongs to The National Institutes of Health, and has Federal founding. More than 8,000 patients with a wide variety of rheumatologic diagnosis receive medical care.

On March 2020, the WHO announced COVID-19 outbreak a pandemic. The first case was registered in Mexico on February 2020. In March 2020, the Mexican Government requested that our Institution should restrict health care to exclusively COVID-19 patients; accordingly, outpatient consultations were, and up to August 2020 still, hold on.

Meanwhile, when possible, the Department of Immunology and Rheumatology has implemented an "on-demand", non-organized patient´s health care, through email and phone contact; nonetheless, and due to the middle-low socioeconomic status of most of our patients and limited technical resources available at our Institution, the attempt has been challenging.

DETAILED DESCRIPTION:
The aim objective of this project is to explore patients perception about access to medical care and to medications, access to communication with their primary rheumatologist and patients risk perception about COVID-19 disease, for this a survey directed (questionnaire locally developed) will apply and to explore how the reintegration at the usual medical care has a positive impact in the patient´s disease activity, patient´s quality of life and psychopathology (depression, anxiety and posttraumatic stress).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a rheumatic disease diagnosis according to their primary rheumatologist who agree to participate

Exclusion Criteria:

* Patients with a not confirmed rheumatic disease
* Patients lost to follow-up from the outpatient for > 1 year period
* Patients with pregnancy plans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the rheumatic diseases outpatients from the National Institute of Medical Sciences and Nutrition that will assist their usual medical care posterior of stopped it during the COVID-19 pandemic.
Sampling Method: Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in the pattern of the usual medical care among the rheumatic disease patients | At study inclusion (The first medical consultation posterior to open the external outpatient's service, post COVID-19 pandemic)
  To determinate the proportion of the rheumatic disease patients affected in their usual medical care during the COVID-19 pandemic in our Institution with the COVID-19 survey (locally development)

SECONDARY OUTCOMES:
Change in the patient's activity disease | In the first medical consultation posterior to open the external outpatient's service (post COVID-19 pandemic) to 6 months follow-up
  Change in the activity disease measured as RAPID-3 of the Rheumatic disease patients in a 6 months follow-up. The results will express with a scale 0 to 30 a > number > disease activity
Change in the patient's activity disease measures by their rheumatologist | In the first medical consultation posterior to open the external outpatient's service (post COVID-19 pandemic) to 6 months follow-up
  Change in the activity disease measured by their rheumatologist (4 questions) of the rheumatic disease patients in a 6 months follow-up. The results will express with 3 categories (without activity, low activity, moderate activity, high activity)
Change in patient´s quality of life | In the first medical consultation posterior to open the external outpatient's service (post COVID-19 pandemic) to 6 months follow-up
  Change in the quality of life measured as WHOQOL-BREF of the Rheumatic disease patients in a 6 months follow-up. The results will express with a scale 0 to 100 a > number > quality of life
Change in patient´s depression and anxiety | In the first medical consultation posterior to open the external outpatient's service (post COVID-19 pandemic) to 6 months follow-up
  Change in the psychopathology measured as DASS-21 instrument (depression and anxiety) of the Rheumatic disease patients in a 6 months follow-up. The results will express with a scale 0 to 8 a cut of point > 8 suggests depression and stress presence, and > 5 suggests anxiety presence
Change in patient´s posttraumatic stress | In the first medical consultation posterior to open the external outpatient's service (post COVID-19 pandemic) to 6 months follow-up
  Change in the psychopathology measured as IER-R (posttraumatic stress) of the Rheumatic disease patients in a 6 months follow-up. The results will express with a scale 0 to 88 a cut of point > 24 would be significant

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pascual-Ramos, Dr., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No